CLINICAL TRIAL: NCT04907487
Title: Évaluation de l'Impact du Compressed Sensing Sur le Signal QSM
Acronym: CS-QSM
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: JSY_2021_13
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: MRI

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SEP: With Multiple Sclerosis as defined by McDonald's revised clinical or radiological spatial and temporal dissemination criteria
  Interventions: Device: MRI
- NO SEP: For patients with an indication to undergo a brain MRI and at low risk of inflammatory CNS disease
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — MRI of routine care includes at least the following sequences:
  * 3D T1 TFE (2 minutes)
  * T2 TSE (2 minutes)
  * 3D FLAIR (3 minutes)
  The sequences added by the research lasting 25 minutes are:
  * SWI QSM 1.0iso 8 echoes (10 minutes)
  * SWI QSM 1.0iso 8 echoes CS 6 (7 minutes)
  * SWI QSM 1.0iso 8 echoes CS 9 (5 minutes)
  * SWI QSM 1.0iso 8 echoes CS 12 (3 minutes)

SUMMARY:
Patients who have agreed to participate in the study will complete the MRI protocol as part of routine care, to which a maximum of four additional 25-minute sequences will be added.

MRI of routine care includes at least the following sequences:

* 3D T1 TFE (2 minutes)
* T2 TSE (2 minutes)
* 3D FLAIR (3 minutes)

The sequences added by the research lasting 25 minutes are:

* SWI QSM 1.0iso 8 echoes (10 minutes)
* SWI QSM 1.0iso 8 echoes CS 6 (7 minutes)
* SWI QSM 1.0iso 8 echoes CS 9 (5 minutes)
* SWI QSM 1.0iso 8 echoes CS 12 (3 minutes)

DETAILED DESCRIPTION:
Patients who have agreed to participate in the study will complete the MRI protocol as part of routine care, to which a maximum of four additional 25-minute sequences will be added.

MRI of routine care includes at least the following sequences:

* 3D T1 TFE (2 minutes)
* T2 TSE (2 minutes)
* 3D FLAIR (3 minutes)

The sequences added by the research lasting 25 minutes are:

* SWI QSM 1.0iso 8 echoes (10 minutes)
* SWI QSM 1.0iso 8 echoes CS 6 (7 minutes)
* SWI QSM 1.0iso 8 echoes CS 9 (5 minutes)
* SWI QSM 1.0iso 8 echoes CS 12 (3 minutes)

ELIGIBILITY:
Inclusion Criteria:

For patients with MS:

* Patient over 18 years old
* Presenting MS defined according to McDonald's revised criteria for spatial and temporal clinical or radiological dissemination [16],
* Should benefit as part of the care of an MRI examination with or without injection of gadolinium
* Express consent to participate in the study
* Affiliate or beneficiary of a social security scheme

For patients with an indication to undergo a brain MRI and at low risk of inflammatory CNS disease:

* Patient over 18 years old
* Should benefit as part of the care of an MRI examination with or without injection of gadolinium
* Express consent to participate in the study
* Affiliate or beneficiary of a social security scheme

Exclusion Criteria:

* For patients with MS:
* Patient benefiting from a legal protection measure
* Pregnant or breastfeeding woman

For patients with an indication to undergo a brain MRI and at low risk of inflammatory CNS disease:

* Patient benefiting from a legal protection measure
* Pregnant or breastfeeding woman
* Patient with inflammatory and / or demyelinating pathology of the CNS

Secondary exclusion criteria :

* Motion artefact not allowing interpretation of images
* Patient who did not perform one of the following sequences: 3D T1 TFE, 3D FLAIR (for MS patients), SWI QSM 1.0iso 8 echoes.

Secondarily excluded patients will be replaced.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two groups of patients will be included as part of this research protocol:
  * Group I: Patients with MS
  * Group II: Patients with an indication to undergo a brain MRI and at low risk of inflammatory CNS pathology, age and gender matched with group I.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-05-14 (Actual)

PRIMARY OUTCOMES:
concordance of QSM signal with and without compressed-sensing in white matter | 1 DAY
  concordance of QSM signal with and without compressed-sensing in white matter

CONTACTS AND LOCATIONS:
Locations (1):
- Hhopital fondation adolphe de rothschild, Paris, Paris, France